CLINICAL TRIAL: NCT01360671
Title: An Open Label Single Arm, Single Centre Study to Investigate the Safety and Efficacy of IV Sildenafil in Neonates With Persistent Pulmonary Hypertension of the Newborn (PPHN)
Brief Title: IV Sildenafil Persistent Pulmonary Hypertension Of The Newborn
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1481294; PPHN MIRROR STUDY
Record Dates: First submitted 2011-05-10; First posted 2011-05-26 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Persistent Pulmonary Hypertension of the Newborn
Keywords: PPHN; persistent pulmonary hypertension of the newborn; sildenafil; iv
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sildenafil (Experimental): iv sildenafil
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — Loading dose of 0.1 mg/kg for 30 minutes followed by maintenance treatment of 0.03 mg/kg.h for up to 14 days

SUMMARY:
To determine the efficacy of iv sildenafil in term and near term infants with PPHN (persistent pulmonary hypertension of the newborn), by measuring the need for inhaled nitric oxide (iNO) or extracorporeal membrane oxygenation (ECMO) compared to a historical control group not treated with sildenafil.

ELIGIBILITY:
Inclusion Criteria:

* Babies < 72 hours old and at least 34 gestational weeks with PPHN or hypoxic respiratory failure associated with idiopathic PPHN, meconium aspiration, sepsis or pneumonia
* Oxygenation index >15 and < 60

Exclusion Criteria:

* Congenital anomaly
* Large left to right intracardiac or ductal shunt
* Already on inhaled nitric oxide

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy - incidence of treatment failure | Day 1-14
Need for inhaled nitric oxide or Extracorporeal membrane oxygenation | Day 1-14

SECONDARY OUTCOMES:
Changes in oxygenation index | 6 & 12 hours
Changes in differential saturation | 6 & 12 hours
Duration of mechanical ventilation | Days 1-14
Time from initiation of sildenafil to inhaled nitric oxide or extracorporeal membrane oxygenation | Days 1-14

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481294&StudyName=IV%20Sildenafil%20Persistent%20Pulmonary%20Hypertension%20Of%20The%20Newborn